CLINICAL TRIAL: NCT06086405
Title: ECMO Braile Biomédica® in COVID-19 Patients Post-market Clinical Trial to Verify the Performance of the ECMO System
Brief Title: ECMO Braile Biomédica® in COVID-19 Patients
Acronym: ECMO_COVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Braile Biomedica Ind. Com. e Repr. Ltda. (Industry)
Responsible Party: Sponsor
Other Study IDs: ECMO COVID
Record Dates: First submitted 2023-10-13; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: COVID-19
Keywords: ECMO; COVID-19; Membrane Oxygenator
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Patients underwent cardiorespiratory support — Patients underwent cardiorespiratory support using the Oxyprime® ECMO Braile Biomédica® Membrane Oxygenator

SUMMARY:
Retrospective data collection to evaluate the gas transfer capacity of the Braile Biomédica® OxyPrime® ECMO BRCoating® Membrane Oxygenator in COVID-19 patients during the pandemic.

DETAILED DESCRIPTION:
Multicenter, retrospective, non-comparative, non-randomized study to assess the clinical performance of the OxyPrime® ECMO BRCoating® Membrane Oxygenator in adult patients with COVID-19

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old, with a previous diagnosis of COVID-19, who were placed on ECMO using the Oxyprime® ECMO Braile Biomédica® Membrane Oxygenator, from March 2020 to July 2022, following the Instructions for Use (IFU) of the products.

Exclusion Criteria:

* Patients without a diagnosis of COVID-19

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients ≥ 18 years old, with a previous diagnosis of COVID-19, who were placed on ECMO using the Oxyprime® ECMO Braile Biomédica® Membrane Oxygenator
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-09-14 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
The effectiveness of the oxygenator in ensuring adequate gas exchange | during the first week of use
  To ensure adequate oxygenation (post-membrane pO2 > 150 mmHg during the first week of use) and CO2 elimination (post-membrane pCO2 < 40 mmHg or pre-membrane pCO2 - post-membrane pCO2 > 10 mmHg)
The effectiveness of the set in ensuring adequate flow to the patient | during the use of extracorporeal membrane oxygenation
  Nominal flow calculated according to weight or body surface area (50 to 80 mL/Kg or 2.4 L/min of body surface area

SECONDARY OUTCOMES:
Rate free of membrane dysfunction | during the use of extracorporeal membrane oxygenation
  percentage of oxygenators free from dysfunction
Need for oxygenator due to dysfunction | during the use of extracorporeal membrane oxygenation
  percentage of oxygenators that needed to be replaced due to dysfunction
Decannulation rate | during the use of extracorporeal membrane oxygenation
  percentage of patients who were decannulated from ECMO
Mortality rate during ECMO use | during the use of extracorporeal membrane oxygenation
  percentage of patients who progressed to mortality during ECMO use
Duration of ECMO system usage | during the use of extracorporeal membrane oxygenation
  Total duration of ECMO use (in days)
Adverse events during extracorporeal membrane oxygenation use | during the use of extracorporeal membrane oxygenation
  percentage of adverse events related to the oxygenator

CONTACTS AND LOCATIONS:
Overall Officials: Vitor S Barzila, Principal Investigator — Hospital Brasília
Locations (1):
- Hospital Brasília, Lago Sul, Brasília - DF, Brazil

IPD SHARING:
Plan to Share IPD: No